CLINICAL TRIAL: NCT03840135
Title: A Multicenter Prospective, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Polyoxidonium, Nasal and Sublingual Spray, 6 mg/ml in Children Aged From 1 to 12 Years With ARI (Acute Respiratory Infection)
Brief Title: Efficacy and Safety of Polyoxidonium, Nasal and Sublingual Spray, 6 mg/ml in Children Aged 1-12 Years With ARI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PoArvi/PhIII_2017
Record Dates: First submitted 2018-11-26; First posted 2019-02-15 (Actual); Results first posted 2020-06-25 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Acute Respiratory Infection
Keywords: ARI, acute respiratory infection
MeSH Terms: interventions — azoximer bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyoxidonium 6 mg/ml (Experimental): Polyoxidonium 6 mg/ml nasal and sublingual spray - 0,15 mg/kg daily - 7 days.
  Interventions: Drug: Polyoxidonium 6 mg/ml
- Placebo (Placebo Comparator): Placebo, nasal and sublingual spray - 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Polyoxidonium 6 mg/ml — Nasal and sublingual spray Polyoxidonium 6 mg/ml will be administered at a dose of 0,15 mg/kg daily for 7 days:
  in children aged from 1 to 2 years - 1 spray sublingually 2 times a day (every 12 hours); in children aged from 2 to 5 years - 1 spray intranasally (in each nasal passage) 2 times a day (every 12 hours; in children aged from 5 to 8 years - 1 spray intranasally (in each nasal passage) 3 times a day (every 8 hours); in children aged from 8 to 12 years - 2 spray intranasally (in each nasal passage) 2 times a day (every 12 hours).
  Other Names: Polyoxidonium, Nasal and Sublingual Spray, 6 mg/ml
  Arms: Polyoxidonium 6 mg/ml
Other: Placebo — Placebo nasal and sublingual spray will be administered for 7 days:
  in children aged from 1 to 2 years - 1 spray sublingually 2 times a day (every 12 hours); in children aged from 2 to 5 years - 1 spray intranasally (in each nasal passage) 2 times a day (every 12 hours; in children aged from 5 to 8 years - 1 spray intranasally (in each nasal passage) 3 times a day (every 8 hours); in children aged from 8 to 12 years - 2 spray intranasally (in each nasal passage) 2 times a day (every 12 hours).
  Other Names: Placebo, Nasal and Sublingual Spray
  Arms: Placebo

SUMMARY:
The purpose of this study is is to demonstrate superiority of Polyoxidonium, nasal and sublingual spray, 6 mg/ml over placebo in children aged from 1 to 12 years with acute respiratory viral infections. This is a multicenter prospective, randomized, double-blind, placebo-controlled, parallel-group phase 3 study.

DETAILED DESCRIPTION:
This is a multicenter prospective, randomized, double-blind, placebo-controlled, parallel-group phase 3 study to evaluate efficacy of Polyoxidonium spray 6 mg/ml on acute respiratory viral infections symptoms in children population. A study will last for 13 days (maximum) for each participant and will include 6 visits: Day 0 (Screening), Day 1, Day 3, Day 5, Day 8 ±1, Day 12 ±1. Express tests will be performed at the screening visit to exclude subjects with influenza or streptococcal infection. All eligible subjects will be treated with Polyoxidonium spray 6 mg/ml or placebo spray for 7 days. Clinical blood and urine tests will be performed at days 0 and 8 ±1. Symptom Assessment Scale (SAS) will be filled in at days 0, 1, 3, 5 and 8 ±1. Integrative Medicine Outcome Scale (IMOS) will be filled in by investigator and a parent/adopter at day 8 ±1. Adverse events information will be collected at days 1, 3, 8 ±1 and 12 ±1.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 1 to 12 years
* Diagnosis of acute respiratory viral infection [International Classification of Diseases (10-th revision) codes: Acute nasopharyngitis [common cold], J02 Acute pharyngitis, J02.9 Acute pharyngitis, unspecified, J04 Acute laryngitis and tracheitis, J04.0 Acute laryngitis, J04.1 Acute tracheitis, J04.2 Acute laryngotracheitis, J06 Acute upper respiratory infections of multiple and unspecified sites, J06.0 Acute laryngopharyngitis, J06.9 Acute upper respiratory infection, unspecified] confirmed by physical examination: axillary temperature ≥ 37,0°C (measured at the moment of physical examination) and Symptoms Assessment Scale total score ≥5 points (not less than 3 of which should be related to ear, or nose, or throat, or upper respiratory tract affection symptoms).
* Less than 24 hours from the onset of disease (first respiratory viral infection symptoms)
* Informed consent signed by parent/adopter, or a child (applicable for children aged > 10 years)

Exclusion Criteria:

* Suspicion on pneumonia, bacterial infection (including meningitis, sepsis, otitis media, sinusitis, sinusitis, urinary tract infection etc.) or a condition that requires antibacterial therapy from the first day of treatment.
* Suspicion on other diseases that may simulate acute respiratory viral infection at the moment of onset (other infectious diseases, flu-like syndrome in system collagen and other diseases).
* Positive express test for influenza or streptococcal infection.
* Clinical signs of serious acute respiratory viral infection, which requires hospitalization (fever ≥ 40°C, sings of airway obstruction, significant hemodynamic or neurological disorders).
* History of primary or secondary immunodeficiency.
* Cancer.
* Acute infectious and non-infectious diseases (except acute respiratory viral infection), exacerbation or decompensation of chronic diseases (diabetes mellitus, infantile cerebral paralysis, cystic fibrosis, primary ciliary dyskinesia, bronchopulmonary dysplasia, malformations of upper respiratory tract,ears, nose, or throat) which may affect an ability of patient to participate in study.
* Saccharase/isomaltase deficiency, fructose intolerance, glucose-galactose malabsorption.
* History of allergy/hypersensitivity to any component of the study drug (including paracetamol, propacetamol hydrochloride).
* Use of protocol-prohibited medications within 1 month prior to study.
* Children, who's parents/adopters may fail to follow the protocol procedures and treatment, in investigator's opinion.
* Participation in other studies within 3 months to screening.
* Pregnancy.
* Any other medical or social condition that may interrupt study participation, in investigator's opinion.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai Dodonov, Study Chair — NPO Petrovax
Locations (11):
- Russia (11):
  - Medical Center "Medical Technology", Saint Petersburg, Leningradskaya Oblast'
  - Medical Center "MedAestheticCentre Laboratory", Saint Petersburg, Leningradskaya Oblast'
  - Medical center "Curator", Saint Petersburg, Leningradskaya Oblast'
  - Children's City Hospital No. 22, Saint Petersburg, Leningradskaya Oblast'
  - Medical center "Korolev Medicine", Naro-Fominsk, Moscow Oblast
  - City Children's Clinical Clinic №5, Perm, Perm Krai
  - Children's City Clinic №4 of the city of Rostov-on-Don, Rostov-on-Don, Rostov Oblast
  - Yaroslavl State Medical University, Yaroslavl, Yaroslavl Oblast
  - Regional Children's Clinical Hospital, Yaroslavl, Yaroslavl Oblast
  - Scientific Clinical Center of Otorhinolaryngology of the Federal Medical and Biological Agency, Moscow
  - Federal state budgetary institution "Research Institute of Influenza" of Ministry of Health of Russia, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garashchenko TI, Karneeva OV, Tarasova GT, Kim IA, Hanferian RA (2020) Efficacy and safety of azoximer bromide (Polyoxidonium) in children aged from 1 to 12 years with ARI: The results of a multicenter prospective, randomized, double-blind, placebo-controlled, parallel-group study. Pediatr Dimensions 5: DOI: 10.15761/PD.1000204.

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyoxidonium 6 mg/ml: Polyoxidonium 6 mg/ml nasal and sublingual spray - 0,15 mg/kg daily - 7 days.
  Polyoxidonium 6 mg/ml: Nasal and sublingual spray Polyoxidonium 6 mg/ml was administered at a dose of 0,15 mg/kg daily for 7 days:
  in children aged from 1 to 2 years - 1 spray 2 times a day sublingually (every 12 hours); in children aged from 2 to 5 years - 1 spray intranasally (in each nasal passage) 2 times a day (every 12 hours); in children aged from 5 to 8 years - 1 spay intranasally (in each nasal passage) 3 times a day (every 8 hours); in children aged from 8 to 12 years - 2 spay intranasally (in each nasal passage) 2 times a day (every 12 hours).
- Placebo: Placebo, nasal and sublingual spray - 7 days.
  Placebo: Placebo nasal and sublingual spray will be administered for 7 days:
  in children aged from 1 to 2 years - 1 spray 2 times a day sublingually (every 12 hours); in children aged from 2 to 5 years - 1 spray intranasally (in each nasal passage) 2 times a day (every 12 hours); in children aged from 5 to 8 years - 1 spay intranasally (in each nasal passage) 3 times a day (every 8 hours); in children aged from 8 to 12 years - 2 spay intranasally (in each nasal passage) 2 times a day (every 12 hours).
Period: Overall Study
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Started | 86 | 86
Completed | 79 | 85
Not Completed | 7 | 1
Not completed — Protocol Violation | 6 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 172 patients were randomized, 8 people dropped out during the trial (due to protocol violations and withdrawal of informed consent). 164 patients completed the study, data from 155 children were accepted for the final analysis (9 patients were excluded from the analysis due to protocol violations).
Groups:
- Polyoxidonium 6 mg/ml: Polyoxidonium 6 mg/ml nasal and sublingual spray - 0,15 mg/kg daily - 7 days.
  Polyoxidonium 6 mg/ml: Nasal and sublingual spray Polyoxidonium 6 mg/ml will be administered at a dose of 0,15 mg/kg daily for 7 days:
  in children aged from 1 to 2 years - 1 sublingual spray 2 times a day (every 12 hours); in children aged from 2 to 5 years - 1 intranasal spray (in each nasal passage) 2 times a day (every 12 hours; in children aged from 5 to 8 years - 1 intranasal spray (in each nasal passage) 3 times a day (every 8 hours); in children aged from 8 to 12 years - 2 intranasal spray (in each nasal passage) 2 times a day (every 12 hours).
- Placebo: Placebo, nasal and sublingual spray - 7 days.
  Placebo: Placebo nasal and sublingual spray will be administered for 7 days:
  in children aged from 1 to 2 years - 1 sublingual spray 2 times a day (every 12 hours); in children aged from 2 to 5 years - 1 intranasal spray (in each nasal passage) 2 times a day (every 12 hours; in children aged from 5 to 8 years - 1 intranasal spray (in each nasal passage) 3 times a day (every 8 hours); in children aged from 8 to 12 years - 2 intranasal spray (in each nasal passage) 2 times a day (every 12 hours).
- Total: Total of all reporting groups
Arm/Group | Polyoxidonium 6 mg/ml | Placebo | Total
Number analyzed (Participants) | 76 | 79 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 76 | 79 | 155
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6 [2 to 8] | 5 [2 to 7] | 5 [2 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 41 | 74
  Male | 43 | 38 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 75 | 78 | 153
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 76 | 79 | 155
Body Mass [Median (Inter-Quartile Range); unit: kg] | 20.85 [14.6 to 30] | 18 [15 to 27] | 19 [14.5 to 28.05]
Body height [Median (Inter-Quartile Range); unit: m] | 1.16 [0.96 to 1.33] | 1.12 [0.98 to 1.29] | 1.13 [0.97 to 1.305]

OUTCOME MEASURES:

1. Primary Outcome: Fever Duration (With a Superiority Cut-off Level δ=-0,52 Days)
Description: Normalization of body temperature (axillary body temperature level ≤ 36,9 °C confirmed by two consecutive measurements (morning-evening/evening-morning)) will be considered as the end of fever
Time Frame: Day 8±1
Measure: Mean (95% Confidence Interval); unit: day
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
day | 2.04 [1.74 to 2.34] | 2.26 [2.03 to 2.50]
Statistical Analysis 1: Comparison: Polyoxidonium 6 mg/ml vs Placebo; The value of δ = -0.52 days was considered as the boundary of superiority. The end of the fever period is considered to have an axillary body temperature of ≤36.9 ° C in two consecutive measurements (morning-evening / evening-morning); Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.6 to 0.16]

2. Secondary Outcome: Changes in Intoxication Symptoms by 3 Day of Treatment Due to Symptom Assessment Scale (SAS)
Description: A total number of patients (NP) without symptoms due to "General intoxication symptoms" domain of the Symptom Assessment Scale (SAS) was evaluated.
  A total number of patients (NP) with mild symptoms due to "General intoxication symptoms" domain of SAS (1 point according SAS) was evaluated.
  A total number of patients (NP) with moderate symptoms due to "General intoxication symptoms" domain of SAS (2 point according SAS) was be evaluated.
  A total number of patients (NP) with severe symptoms due to "General intoxication symptoms" domain of SAS (3 point according SAS) was evaluated.
  Domain "General intoxication symptoms" includes the following symptoms:
  * altered/decreased activity;
  * altered appetite;
  * unhealthy appearance;
  * altered or interrupted sleep.
  Each symptom may be graded by the following points:
  * 0 points - absent;
  * 1 point - mild;
  * 2 points - moderate;
  * 3 points - severe.
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
Participants
  NP without altered/decreased activity day 0 | 14 | 11
  NP with mild altered/decreased activity day 0 | 40 | 51
  NP with moderate altered/decreased activity day 0 | 22 | 17
  NP with severe altered/decreased activity day 0 | 0 | 0
  NP without altered/decreased activity day 3 | 52 | 46
  NP with mild altered/decreased activity day 3 | 23 | 33
  NP with moderate altered/decreased activity day 3 | 1 | 0
  NP with severe altered/decreased activity day 3 | 0 | 0
  NP without altered appetite day 0 | 9 | 10
  NP with mild altered appetite day 0 | 35 | 44
  NP with moderate altered appetite day 0 | 31 | 25
  NP with severe altered appetite day 0 | 1 | 0
  NP without altered appetite day 3 | 54 | 50
  NP with mild altered appetite day 3 | 18 | 27
  NP with moderate altered appetite day 3 | 4 | 2
  NP with severe altered appetite day 3 | 0 | 0
  NP without unhealthy appearance day 0 | 8 | 6
  NP with mild unhealthy appearance day 0 | 50 | 56
  NP with moderate unhealthy appearance day 0 | 18 | 17
  NP with severe mild unhealthy appearance day 0 | 0 | 0
  NP without unhealthy appearance day 3 | 59 | 49
  NP with mild unhealthy appearance day 3 | 16 | 30
  NP with moderate unhealthy appearance day 3 | 1 | 0
  NP with severe unhealthy appearance day 3 | 0 | 0
  NP without altered or interrupted sleep day 0 | 40 | 46
  NP with mild altered or interrupted sleep day 0 | 23 | 27
  NP with moderate altered or interrupt. sleep day 0 | 13 | 6
  NP with severe altered or interrupt. sleep day 0 | 0 | 0
  NP without altered or interrupted sleep day 3 | 73 | 71
  NP with mild altered or interrupted sleep day 3 | 3 | 6
  NP with moderate altered or interrupt. sleep day 3 | 0 | 2
  NP with severe altered or interrupt. sleep day 3 | 0 | 0
Statistical Analysis 1: Comparison: Polyoxidonium 6 mg/ml vs Placebo; Test type: Superiority; p < 0.05, χ2 Pearson criterion

3. Secondary Outcome: Number of Patients (NP) Without Nasal Discharge Symptom by 3 and 5 Day of Treatment, Number of Patients (NP) With Mild/Moderate/Severe Nasal Discharge Symptom by 3 and 5 Day of Treatment
Description: Each symptom was graded by the following points:
  * 0 points - absent;
  * 1 point - mild;
  * 2 points - moderate;
  * 3 points - severe. Number of patients (NP) without nasal discharge symptom by 3 and 5 day of treatment (score on the scale 0 point), Number of patients (NP) with mild nasal discharge symptom by 3 and 5 day of treatment (score on the scale 1 points) Number of patients (NP) with moderate nasal discharge symptom by 3 and 5 day of treatment (score on the scale 2 points) Number of patients (NP) with severe nasal discharge symptom by 3 and 5 day of treatment (score on the scale 3 points)
Time Frame: Day 3, Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
Participants
  Day 0: NP without nasal discharge symptom | 9 | 12
  Day 0: NP with mild nasal discharge symptom | 19 | 20
  Day 0: NP with moderate nasal discharge symptom | 46 | 43
  Day 0: NP with severe nasal discharge symptom | 2 | 4
  Day 3: NP without nasal discharge symptom | 26 | 13
  Day 3: NP with mild nasal discharge symptom | 30 | 37
  Day 3: NP with moderate nasal discharge symptom | 20 | 29
  Day 3: NP with severe nasal discharge symptom | 0 | 0
  Day 5: NP without nasal discharge symptom | 40 | 24
  Day 5: NP with mild nasal discharge symptom | 29 | 38
  Day 5: NP with moderate nasal discharge symptom | 7 | 17
  Day 5: NP with severe nasal discharge symptom | 0 | 0
Statistical Analysis 1: Comparison: Polyoxidonium 6 mg/ml vs Placebo; Test type: Superiority; p < 0.05, χ2 Pearson criterion

4. Secondary Outcome: Score on Symptoms: Nasal Discharge and Nasal Congestion/Impaired Nasal Airflow Due to Symptom Assessment Scale by 3 and 5 Day of Treatment
Description: Each symptom was graded by the following points:
  * 0 points - absent;
  * 1 point - mild;
  * 2 points - moderate;
  * 3 points - severe. The higher scores mean worse outcome. The maximum score is 3 points, the minimum score is 0 points.
Time Frame: Day 3, Day 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
score on a scale
  nasal discharge day 0 | 2 [1 to 2] | 2 [1 to 2]
  nasal discharge by day 3 | 1 [0 to 2] | 1 [1 to 2]
  nasal discharge by day 5 | 0 [0 to 1] | 1 [0 to 1]
  nasal congestion/impaired nasal airflow by day 0 | 2 [2 to 2] | 2 [1 to 2]
  nasal congestion/impaired nasal airflow by day 3 | 1 [0 to 1] | 1 [1 to 2]
  nasal congestion/impaired nasal airflow by day 5 | 0 [0 to 1] | 1 [0 to 1]
Statistical Analysis 1: Comparison: Polyoxidonium 6 mg/ml vs Placebo; Test type: Superiority; p < 0.05, χ2 Pearson criterion

5. Secondary Outcome: Total Score on Symptom Assessment Scale by 3 and 5 Day of Treatment
Description: Symptom Assessment Scale (SAS) consists of 3 domains:
  1. Domain "General intoxication symptoms" (altered/increased activity/dysfunctional behavior; altered appetite or food refusal; unhealthy or alter from common appearance; altered or interrupted sleep);
  2. "Nose symptoms" (nasal discharge; nasal congestion/impaired nasal airflow; sneezing);
  3. "Throat and thoracic symptoms" (hoarseness; sore throat; cough).
  Each symptom may be graded by the following points:
  * 0 points - absent;
  * 1 point - mild;
  * 2 points - moderate;
  * 3 points - severe. The higher scores mean a worse outcome. The total score is the sum of points of each symptom graded in Symptom Assessment Scale. The maximum possible value of the total score is 30 points, the minimum possible value of the total score is 0 points.
Time Frame: Day 3, Day 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
score on a scale
  Day 0 | 11 [8 to 14] | 10 [8 to 13]
  Day 3 | 4.00 [2.00 to 6.00] | 5.00 [3.00 to 7.00]
  Day 5 | 1.00 [0 to 4] | 3.00 [1 to 5]
Statistical Analysis 1: Comparison: Polyoxidonium 6 mg/ml vs Placebo; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Assessment of Treatment Results With Integrative Medicine Outcome Scale (IMOS) Performed by Investigator
Description: Integrative Medicine Outcome Scale (IMOS) is used to assess treatment efficacy and has the following gradations of health condition:
  0 points - absolute recovery;
  1. point - significant improvement;
  2. points - slight to moderate improvement;
  3. points - unchanged;
  4. points - decline. The results is presented in number of patients with 0 points (absolute recovery), number of patients with 1 points (significant improvement), number of patients with 2 points (slight to moderate improvement), number of patients with 3 points (unchanged), number ot patients with 4 points (decline) by day 8 according IMOS.
Time Frame: Day 8±1
Measure: Count of Participants; unit: Participants
Groups:
- Polyoxidonium 6 mg/ml: Polyoxidonium 6 mg/ml nasal and sublingual spray - 0,15 mg/kg daily - 7 days.
  Polyoxidonium 6 mg/ml: Nasal and sublingual spray Polyoxidonium 6 mg/ml will be administered at a dose of 0,15 mg/kg daily for 7 days:
  in children aged from 1 to 2 years - 1 spray sublingually 2 times a day (every 12 hours); in children aged from 2 to 5 years - 1 spray intranasally (in each nasal passage) 2 times a day (every 12 hours; in children aged from 5 to 8 years - 1 spray intranasally (in each nasal passage) 3 times a day (every 8 hours); in children aged from 8 to 12 years - 2 spray intranasally (in each nasal passage) 2 times a day (every 12 hours).
- Placebo: Placebo, nasal and sublingual spray - 7 days.
  Placebo: Placebo nasal and sublingual spray will be administered for 7 days:
  in children aged from 1 to 2 years - 1 spray sublingually 2 times a day (every 12 hours); in children aged from 2 to 5 years - 1 spray intranasally (in each nasal passage) 2 times a day (every 12 hours; in children aged from 5 to 8 years - 1 spray intranasally (in each nasal passage) 3 times a day (every 8 hours); in children aged from 8 to 12 years - 2 spray intranasally (in each nasal passage) 2 times a day (every 12 hours).
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
Participants
  absolute recovery | 62 | 60
  significant improvement | 12 | 14
  slight to moderate improvement | 2 | 4
  unchanged | 0 | 1
  decline | 0 | 0
Statistical Analysis 1: Comparison: Polyoxidonium 6 mg/ml vs Placebo; Test type: Superiority; p < 0.05, χ2 Pearson criterion

7. Secondary Outcome: Assessment of Treatment Results With Integrative Medicine Outcome Scale (IMOS) Performed by Parent/Adopter
Description: as for outcome 6
Time Frame: Day 8±1
Measure: Count of Participants; unit: Participants
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
Participants
  absolute recovery | 41 | 35
  significant improvement | 30 | 30
  slight to moderate improvement | 5 | 9
  unchanged | 0 | 5
  decline | 0 | 0
Statistical Analysis 1: Comparison: Polyoxidonium 6 mg/ml vs Placebo; Test type: Superiority; p < 0.05, χ2 Pearson criterion

8. Secondary Outcome: Number of Cases of Antifebrile Agents Use
Description: Number of cases of the antipyretic product (paracetamol) consumption for the entire study period
Time Frame: Day 8±1
Measure: Count of Participants; unit: Participants
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
Participants | 8 | 10

9. Secondary Outcome: Number of Patients Discontinued From the Study Due to Requirement for Antibacterial Therapy
Description: Number of patients who discontinued from the study due to requirement for antibacterial therapy
Time Frame: Day 8±1
Measure: Count of Participants; unit: Participants
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
Participants | 0 | 0

10. Secondary Outcome: Number of Patients With Normalization of Body Temperature by 5 Day of Treatment
Description: Axillary body temperature level ≤ 36,9 °C confirmed by two consecutive measurements (morning-evening/evening-morning will be considered as normalization of body temperature
Time Frame: Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
Participants | 73 | 76
Statistical Analysis 1: Comparison: Polyoxidonium 6 mg/ml vs Placebo; Test type: Superiority; p < 0.05, Fisher Exact

11. Secondary Outcome: Number of Patients With Clinical Improvement (Symptom Assessment Scale Total Score ≤ 3) by 5 Day of Treatment
Description: Symptom Assessment Scale (SAS) consists of 3 domains:
  1. Domain "General intoxication symptoms" (altered/increased activity/dysfunctional behavior; altered appetite or food refusal; unhealthy or alter from common appearance; altered or interrupted sleep);
  2. "Nose symptoms" (nasal discharge; nasal congestion; impaired nasal airflow; sneezing);
  3. "Throat and thoracic symptoms" (hoarseness; sore throat; cough). The higher scores mean a worse outcome. The total score is the sum of points of each symptom graded in Symptom Assessment Scale. The maximum possible value of the total score is 30 points, the minimum possible value of the total score is 0 points.
  Each symptom may be graded by the following points:
  * 0 points - absent;
  * 1 point - mild;
  * 2 points - moderate;
  * 3 points - severe.
Time Frame: Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
Number analyzed (Participants) | 76 | 79
Participants | 56 | 51
Statistical Analysis 1: Comparison: Polyoxidonium 6 mg/ml vs Placebo; Test type: Superiority; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 12±1 days
Description: Among 172 randomized patients, 2 patients did not take the study drug for reasons of non-compliance with inclusion criterion No. 3 and withdrawal of informed consent, respectively. Thus, the safety analysis included data from 170 patients (84 in the study drug group and 86 in the comparison drug group) who were included in the study and took the drug at least once.
Arm/Group | Polyoxidonium 6 mg/ml | Placebo
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/86
Other Adverse Events (participants affected / at risk) | 1/84 | 6/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyoxidonium 6 mg/ml (N=84) | Placebo (N=86)
acute catarrhal otitis media on the left (Ear and labyrinth disorders) | 1 (1) | 0 (0)
acute purulent otitis media on the left (Ear and labyrinth disorders) | 0 (0) | 1 (1)
loose stool (Gastrointestinal disorders) | 0 (0) | 2 (2)
acute otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
nose bleed (Investigations) | 0 (0) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT03840135/Prot_SAP_ICF_000.pdf